CLINICAL TRIAL: NCT05247762
Title: Effect of Acupuncture on Visual Acuity and Visual Field in Patients With Primary Open-angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH110-REC2-225
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Primary Open-angle Glaucoma
Keywords: Acupuncture
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham acupuncture group (Sham Comparator): Use Wangbuliu Xingzi Paste on the skin, once a week, once for 20 minutes, for 24 weeks.
  Interventions: Device: Acupuncture
- Acupuncture group (Experimental): Use stainless steel needles on the skin, once a week, once for 20 minutes, for 24 consecutive weeks.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — The stainless steel needles are used to insert into the two points of Jingming and the Qiuhou, and der-qi, once a week, once for 20 minutes, for 24 consecutive weeks.

SUMMARY:
The goal of this clinical trial is to test the therapeutic effect of acupuncture at the Jingming and the Qiuhou acupoints on the visual acuity and visual field in patients with primary open-angle glaucoma.

Participants will get acupuncture or Wangbuliu Xingzi Paste (sham acupuncture) on both sides of the Jingming and the Qiuhou, once a week, once for 20 minutes, for 24 weeks.

Researchers will compare acupuncture group and sham acupuncture group to see if the visual acuity, visual field, intraocular pressure, optic nerve fiber layer thickness, serum homocysteine concentration, and scores on the WHOQOL-REF (Taiwan version) scale would be improved.

DETAILED DESCRIPTION:
Glaucoma is a syndrome. The long-term increase in intraocular pressure eventually leads to visual field defect and blindness. Lowering the intraocular pressure in patients with glaucoma is considered to be the most effective way to treat glaucoma. Many studies believe that both blood circulation around the eyes and increased intraocular pressure play a critical role in glaucoma. Some studies have shown that acupuncture can adjust intraocular pressure and improve optic nerve activity, as well as increase blood flow of the eye fundus. Jingming (BL1) can communicate yin and yang, nourish and improve eyesight, and Qiuhou (EX-HN7) can promote qi and blood circulation, and improve vision. The results of our previous research found that acupuncture or electroacupuncture can reduce the intraocular pressure in patients with glaucoma. Therefore, the purpose of this study is to assess the therapeutic effect of acupuncture at the Jingming and the Qiuhou acupoints on the visual acuity and visual field in patients with primary open-angle glaucoma. This study designed a randomized, single-blind, controlled clinical trial. A total of 40 patients with primary open-angle glaucoma were randomly divided into two groups equally as follows: 1) Sham acupuncture group: Only use Wangbuliu Xingzi Paste on the skin on the acupoints on both sides of the Jingming and the Qiuhou, once a week, once for 20 minutes, for 24 weeks; 2) Acupuncture group: The method is the same as the sham acupuncture group, but the stainless steel needles are used to insert into the two points of Jingming and the Qiuhou, and der-qi, once a week, once for 20 minutes, for 24 consecutive weeks. The main assessment is visual acuity and visual field; the secondary assessment includes intraocular pressure, optic nerve fiber layer thickness, serum homocysteine concentration, and changes in scores on the WHOQOL-REF (Taiwan version) scale.

It is expected that acupuncture intervention can improve the visual acuity and visual field in patients with glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Open-angle glaucoma diagnosis at least 3 months previously.
2. Use of one or no intraocular hypotensive drugs.
3. There is no evidence of other eye diseases other than glaucoma.
4. Clear consciousness that enabled the participant to sign the informed consent form and cooperate with the trial procedure.

Exclusion Criteria:

1. Comorbidity with other chronic diseases, such as hypertension and diabetes, and taking multiple drugs.
2. Laser surgery for either glaucoma or myopia.
3. Pregnancy or lactation.
4. Intolerance to acupuncture treatment.
5. Allergy to acupuncture needles.
6. Refusal to sign the informed consent form.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
visual acuity | 24 weeks
  Primary outcome measure was the changes of visual acuity
visual field | 24 weeks
  Primary outcome measure was the changes of visual field

SECONDARY OUTCOMES:
intraocular pressure | 24 weeks
  Secondary outcome measure was the changes of intraocular pressure
optic nerve fiber layer thickness | 24 weeks
  Secondary outcome measure was the changes of optic nerve fiber layer thickness
serum homocysteine concentration | 24 weeks
  Secondary outcome measure was the changes of serum homocysteine concentration
the World Health Organization Quality of Life brief (Taiwan version) scale | 24 weeks
  Secondary outcome measure was the changes of the World Health Organization Quality of Life brief (Taiwan version) scale. The score is between 0-140, and higher score means better life quality.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Liang Hsieh, Ph.D, Principal Investigator — Professor
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan

IPD SHARING:
Plan to Share IPD: No